CLINICAL TRIAL: NCT05184348
Title: Plexin B2 Gene Expression and Polymorphisms in Psoriasis : Relation to NB-UVB, Acitretin and Combined Therapy
Brief Title: Plexin B2 Gene Expression and Polymorphisms in Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ebtehal alaa el Dean kotop Mohamed, MD, Assitant lecturer of Dermatology, Venereology & Andrology, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ebtehal Mohamed
Record Dates: First submitted 2021-11-23; First posted 2022-01-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Acitretin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Narrow band Ultraviolet B phototherapy group (Active Comparator): Patients will be treated with Narrow band Ultraviolet B phototherapy 3 sessions weekly for 3 months with maximum dose of 1400 mJ/cm2.
  Interventions: Radiation: Narrow band Ultraviolet B phototherapy group
- Acitretin group (Active Comparator): Patients will be treated with Acitretin in dose of 0.5-1 mg per kg per day orally for 3 months
  Interventions: Drug: Acitretin group
- Acitretin plus Narrow band Ultraviolet B phototherapy group (Active Comparator): Patients will be treated with Acitretin in dose of 0.5-1 mg per kg per day orally plus NB-UVB phototherapy 3 sessions weekly for 3 months with maximum dose 1400 mJ/cm2.
  Interventions: Combination Product: Acitretin plus Narrow band Ultraviolet B phototherapy group
- Control group (No Intervention): 30 healthy individuals un related , age, sex , BMI matched with volunteers.

INTERVENTIONS:
Radiation: Narrow band Ultraviolet B phototherapy group — 3 sessions weekly for 3 months with maximum dose 1400 mJ/cm2.
  Other Names: NB-UVB
  Arms: Narrow band Ultraviolet B phototherapy group
Drug: Acitretin group — dose of 0.5-1 mg per kg per day orally for 3 month.
  Arms: Acitretin group
Combination Product: Acitretin plus Narrow band Ultraviolet B phototherapy group — Acitretin in dose of 0.5-1 mg per kg per day orally plus Narrow band Ultraviolet B phototherapy 3 sessions weekly for 3 months with maximum dose 1400 mJ/cm2.
  Arms: Acitretin plus Narrow band Ultraviolet B phototherapy group

SUMMARY:
Patients will be randomly assigned (1:1:1 ) either to ; NB-UVB photo-therapy alone , Acitretin therapy alone or NB-UVB photo-therapy combined with Acitretin therapy randomization will be done by closed envelopes . investigator will be blinded to study drug assignment , while patients and data interpreter will not be masked to study drug assignment.

DETAILED DESCRIPTION:
Study Setting: Qena University Hospital, Department of Dermatology ,Venereology& Andrology.

Study subjects: the study will include psoriasis Vulgaris patients who Come to the out patients dermatologic clinic and matching inclusion & exclusion criteria as follow, from 9/2021 up to 3/2023 and then patients will be divided to each group equally as follow:

Group 1: Patients will be treated with NB-UVB phototherapy 3 sessions weekly for 3 months with maximum dose of 1400 mJ/cm2.

Group 2: Patients will be treated with Acitretin in dose of 0.5-1 mg per kg per day orally for 3 months Group 3: Patients will be treated with Acitretin in dose of 0.5-1 mg per kg per day orally plus NB-UVB phototherapy 3 sessions weekly for 3 months with maximum dose 1400 mJ/cm2.

Group 4: 30 healthy individuals un related , age, sex , BMI matched with volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes. Diagnosed clinically with moderate to severe Psoriasis Vulgaris.
* patients able to swallow tablet and receive Narrow band Ultraviolet B phototherapy without any contraindication

Exclusion Criteria:

Pregnancy , lactation & women intent to become pregnant within 3 year after discontinuation of acitretin Patients with Hyperlipidemia Patients with mental problems and depression Patients with a history of malignancies, renal & liver diseases. Patients with a history of any inflammatory diseases as atopic dermatitis , asthma ulcerative colitis ) and Crohn's disease Patients received NB-UVB phototherapy in the last 6 months. Patients treated with methotrexate or biologic agents and any systemic treatment of psoriasis.

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Improve the prognosis of patients with psoriasis Vulgaris | 3 month
  detect the effect of Acitretin alone and Narrow band Ultraviolet B phototherapy alone versus combined therapy on genetic mutation and level of plexin b2 in patients with psoriasis Vulgaris

SECONDARY OUTCOMES:
Improve the clinical out comes of patients with psoriasis Vulgaris | 12 month
  detect the effect of Acitretin alone and Narrow band Ultraviolet B phototherapy alone versus combined therapy on clinical out comes and PASI score of patients with psoriasis Vulgaris

CONTACTS AND LOCATIONS:
Overall Officials: Eisa Hegazy, Prof., Study Chair — Faculty of Medicine, South Valley University, Egypt
Locations (1):
- Faculty of Medicine , South Valley University, Qina, Egypt